CLINICAL TRIAL: NCT04578587
Title: Reliability of Hand Held Dynamometer for Assessing Isometric Lumbar Muscle Strength in Asymptomatic Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fahad Tanveer (Other)
Responsible Party: Sponsor-Investigator, Fahad Tanveer, Assistant Professor, University of Lahore
Organization: University of Lahore (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: IRB-UOL-FAHS/690/2020
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: Reliability; Lumbar region; Muscle strength dynamometer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Rater 1 (Active Comparator): Rater 1
  Interventions: Device: MicroFET 2
- Rater 2 (Active Comparator): Rater 2
  Interventions: Device: MicroFET 2

INTERVENTIONS:
Device: MicroFET 2 — Lumbar Flexor and Extensor Strength Measurement

SUMMARY:
To determine intra-rater and inter-rater reliability of hand held dynamometer for assessing isometric lumbar

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants given informed consent underwent a 1-week screening period to determine eligibility for study entry. Two raters assessed isometric strength of lumbar flexor and extensor muscles, by a hand-held dynamometer. Strength was measured and recorded by each of the two raters and re-assessed after a week.

ELIGIBILITY:
Inclusion Criteria:

* age between twenty one to twenty five years

Exclusion Criteria:

* subjects with the history of acute, subacute or chronic low back pain, history of trauma, neurological disorders, spinal surgery, lumbar spine pathology were excluded.

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Hand held dynamometer | 2 Weeks
  Muscle Strength

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No